CLINICAL TRIAL: NCT03322059
Title: Randomized Trial of Charity-based Incentives to Increase Physical Activity Among Cancer Survivors
Brief Title: Evaluating Whether Charity Incentives Motive Cancer Survivors to Increase Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Sarah K Keadle, Assistant Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSCA111
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cancer; Physical Activity; Incentives
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The core intervention will include educational materials, access to a basic smartphone app and a Fitbit.
  Participants will receive a weekly email with a step goal that will increase 10% beyond the previous weeks values.
  Interventions: Behavioral: Control
- Intervention (Experimental): The core intervention will include educational materials, access to a basic smartphone app and a Fitbit. Participants will receive a weekly email with a step goal that will increase 10% beyond the previous weeks values.
  Participants will be in the form of a charitable donation in their name to a cancer charity.
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — Participants will receive a fitbit and lifestyle counseling to increase steps. Weekly newsletter for first 6 weeks, bi-weekly for remaining weeks with behavioral content designed to increase physical activity (e.g., barriers, SMART goals). They will also receive a donation to a cancer charity of their choice if they meet daily step goals.
  Other Names: Fitbit+incentives
  Arms: Intervention
Behavioral: Control — Participants will receive a fitbit and lifestyle counseling to increase steps. Weekly newsletter for first 6 weeks, bi-weekly for remaining weeks with behavioral content designed to increase physical activity (e.g., barriers, SMART goals).
  Other Names: Fitbit-only
  Arms: Control

SUMMARY:
The investigators propose to examine whether linking daily activity with charity-based incentives motivates cancer survivors to initiate and maintain physical activity. Linking daily physical activity goals with a cancer specific charity incentive may provide a uniquely salient motivator that promotes increased physical activity among cancer survivors. The investigators will examine whether using activity monitors in combination with charitable incentives leads to greater increases in physical activity compared to activity monitors alone. Target participants includes cancer survivors who are not already active. Physical activity (e.g., steps per day, time in moderate-intensity activity) will be examined at baseline and following a 12-week intervention period using an activPAL accelerometer. After the baseline assessment, both groups will receive a fitbit monitor and informational material designed to increase physical activity. Participants in the fitbit+charity group will have donations made in their name to a cancer charity if they meet daily step goals. Physical activity levels will be monitored using the fitbit device for 6-weeks following the formal intervention period.

DETAILED DESCRIPTION:
The study is a Randomized Controlled Trial (RCT) of a 12-week physical activity intervention. Fifty cancer survivors will be recruited and allocated to one of two research arms: Fitbit+Only Group or Fitbit+Charity Incentives Group. Participants in both intervention arms will be asked to track their physical activities using Fitbit One, an activity monitor that monitors steps and physical activity and will receive basic educational materials about increasing physical activity. Those in the Fitbit+charity incentives Group will raise money for cancer charities if they meet weekly step targets.

The key outcome variable of the RCT is steps as measured by an activPAL accelerometer. Data will be collected at baseline and 12-weeks. Fitbit data will also be collected for the duration of the 12-week intervention and for 6-weeks following the end of the intervention period to have an initial examination of behavior change maintenance (total 18-weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years and <50 y, with diagnosed Adolescent or Young Adult cancer (diagnosed between 15-39y of age);
2. ≥ 6 months post-cancer treatment
3. English speaking
4. Participate in <60 minutes of MVPA/week
5. Own a smartphone
6. Have access to computer
7. Participants must also pass a physical activity readiness questionnaire or receive medical clearance from their primary care physician or oncologist.

Exclusion Criteria:

1. Joint, cardiovascular, or respiratory problem(s) precluding physical activity
2. Metastatic disease
3. Planned elective surgery or pregnancy during intervention/follow-up that would interfere with participation (e.g., breast reconstructive surgery).
4. Already using a wearable device >5 days per week

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Daily steps | 12 weeks - change from baseline to 12 weeks
  Daily steps as measured by activPAL

SECONDARY OUTCOMES:
Participant retention | 12 weeks
  Proportion of participants retained of those randomized
Intervention Reach | Baseline
  Proportion of individuals who agree to participate of those who express an interest in participation
Step goal adherence | 1-12 weeks
  Proportion of weeks meeting physical activity goal as measured by fitbit
Daily Steps | baseline to 12 weeks
  Daily Steps as Measured by Fitbit
Sleep | baseline to 12 weeks
  Sleep as Measured by Fitbit
Sedentary time | Change from baseline to 12 weeks
  Sedentary time as Measured by activPAL activity monitor
Standing time | Change from baseline to 12 weeks
  Standing time as Measured by activPAL
Stepping time | Change from baseline to 12 weeks
  Stepping time as Measured by activPAL
Moderate-vigorous intensity physical activity (MVPA) time | Change from baseline to 12 weeks
  MVPA time as Measured by activPAL
Sedentary breaks/patterns | Change from baseline to 12 weeks
  Sedentary breaks/patterns as Measured by activPAL
Fatigue | Change from baseline to 12 weeks
  Patient-Reported Outcomes Measurement Information System Fatigue Short Form 8a (Total Score range 8-40). higher score is more fatigue.
Physical Function | Change from baseline to 12 weeks
  Patient-Reported Outcomes Measurement Information System Physical Function Short Form 20a. Total score (range 20-100). Higher score is worse physical function
Depression | Change from baseline to 12 weeks
  Patient-Reported Outcomes Measurement Information System Depression Short Form 8a. Total score range 8-40. Higher score is more depressed.
Attitudes Toward Charitable Giving | Change from baseline to 12 weeks
  Attitudes Toward Charitable Giving Scale. Total of 20 questions with scores from 1-5, there are five domains higher score is more of a particular attitude. 1.) Inefficiency of Charitable Giving 2.) Efficiency of Charitable Giving 3.) Cynical Giving 4.) Altruistic Giving 5.) Purpose of Charity
Behavioral Regulation in Exercise Questionnaire | Change from baseline to 12 weeks
  Behavioral Regulation in Exercise Questionnaire -3. Contains 6 subscales Amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, intrinsic regulation, each range from 0-16, higher values indicate more motivation in that domain.
Barriers Self-efficacy Scale | Change from baseline to 12 weeks
  Barriers Self-efficacy Scale. 15 items, total score range 0-1500. Higher indicated more self-efficacy
Physical Activity Enjoyment | Change from baseline to 12 weeks
  Physical Activity Enjoyment Scale. 18-item scale with 7-point bipolar rating. Total score range 18-126. Higher scores reflect greater levels of enjoyment.
Pittsburg Sleep Quality Questionnaire | Change from baseline to 12 weeks
  Pittsburg Sleep Quality Questionnaire. Total score. Greater than 5 indicated poor sleep quality.
Exercise Self-efficacy Scale | Change from baseline to 12 weeks
  Exercise Self-efficacy Scale. 6 items total score. Range 0-600, higher is more self-efficacy
Intervention Maintenance | 12-18 weeks
  % of weeks adhered to step goal as measured by fitbit during 6-week follow-up period
Duration wore Fitbit | 12-18 weeks
  Duration wore Fitbit during during 6-week follow-up period
Exercise outcome expectations | Change from baseline to 12 weeks
  Multidimensional Outcome Expectations for Exercise Scale. Total score (range 15-75), higher score means more multidimensional outcome expectations.
Sleep disturbance | Change from baseline to 12 weeks
  Patient-Reported Outcomes Measurement Information System Sleep Disturbance Form. Total score range 8-40. Higher score is more disturbance.
Exercise Goal Setting | Change from baseline to 12 weeks
  10-item total score. Ranged from 10 to 50, higher score means more goal setting. Exercise Goal-Setting Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

REFERENCES:
- [Derived] Keadle SK, Meuter L, Phelan S, Phillips SM. Charity-based incentives motivate young adult cancer survivors to increase physical activity: a pilot randomized clinical trial. J Behav Med. 2021 Oct;44(5):682-693. doi: 10.1007/s10865-021-00218-w. Epub 2021 Apr 7. PMID 33825070